CLINICAL TRIAL: NCT06004700
Title: Improving Virtual Care of Arthritis: Integrating a Smartphone App Into the EHR for Improved Timeliness of Visits (An Electronic Health Record Integrated Application for Psoriatic Arthritis Patient Reported Outcomes) (RAPID-PsA)
Brief Title: Improving Virtual Care of Arthritis: Integrating a Smartphone App Into the EHR for Improved Timeliness of Visits
Acronym: RAPID-PsA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Daniel H. Solomon, M.D.,MPH, Professor of Medicine, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021P000790
Record Dates: First submitted 2023-08-07; First posted 2023-08-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Arthritis; Psoriatic Arthritis
Keywords: Arthritis; Psoriatic Arthritis; Mobile Health
MeSH Terms: conditions — Arthritis; Arthritis, Psoriatic

STUDY DESIGN:
Masking Description: A matched control group will be enrolled from medical records. The data analyst will be blinded to the treatment assignment (i.e., app intervention or matched controls)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Application (Experimental): This arm of the study will contain half the study population after randomization. The participants in this arm will receive the EHR integrated app and follow a 12-month interrupted time series analysis (ITSA) design.
  n = 260
  Interventions: Other: Mobile Application
- Controls (No Intervention): This arm of the study will contain half the study population after randomization. The participants in this arm will be from the same rheumatologists as the experimental participants and will be used as concurrent controls by accessing their data on visits from the EHR during the same time period.
  n = 260

INTERVENTIONS:
Other: Mobile Application — The current app contains a disease activity questionnaire, a mood scale, a sleep scale, a pain scale, and a functional status scale. The app triggers a brief set of questions each day and allows patients to answer them within 24 hours.
  Arms: Mobile Application

SUMMARY:
The overall objective of this proposal is to test version 3.0 of the Arthritis smartphone app in a 12-month interrupted time series analysis (ITSA) design which will allow us to observe possible differences in visit frequency between the pre-and post-intervention periods as well as between the concurrent control group and those who receive the app. Our central hypothesis is that introduction of the app will reduce visit numbers per month in the group receiving the app, compared with a concurrent control group.

DETAILED DESCRIPTION:
Aim 1: To integrate an app for PsA into the EHR. In current work, user-centered design helped develop an EHR integrated PRO-based app for RA. The roll out of the app has been successful and the investigators now want to expand to focus on integration of a similar app for PsA. The app will use similar PROs, adding in a patient global VAS, as well as a brief psoriasis symptom checklist. The PROMIS Function Short Form, PROMIS Fatigue Short Form, PROMIS Pain Short Form, and the PsAID-12 will be assessed. As well, the Q&A function will be modified to focus on PsA, allowing one to monitor symptom changes for patients using various PsA treatments, focusing on guselkumab, infliximab, golimumab, and ustekinumab. Aim 1 is required for the app testing in Aim 2.

Aim 2: To conduct a single arm interrupted time series of the EHR-integrated PRO app for PsA to assess whether it improves the timeliness of care. After integrating the app into the EHR, the investigators will recruit 100 patients who use one of the following agents: guselkumab, infliximab, golimumab, or ustekinumab. The goal will be to determine whether the app improves visit timeliness. Timeliness will be defined as an increase in the percent of visits with therapeutic changes over a 9-month trial period. A secondary outcome will assess PROs and visit satisfaction. The app allows patients to remotely transmit PRO data to their care team. Patients with very active disease between visits may consider a visit earlier than scheduled. The investigators hypothesize that during the intervention period with app use, patients will experience improved timeliness of PsA care when compared with the 9 months prior to the app use, while maintaining patient-reported clinical outcomes.

Data collection will occur via three methods. First, RA/PsA patients will provide answers to the survey questions through the app on their smartphones or tablets and the ePRO data can be viewed in an administrative dashboard. Second, the app will push an in-basket message to rheumatologists letting them know 1 week before a patient visit that there are ePRO data in Epic to be viewed. If symptoms reach a threshold suggesting poor disease control, then prior to 1 week before the visit the app will send an in-basket message to the rheumatologists letting them know to review patient data to consider an earlier visit. On the other hand, if the ePRO data suggests stable symptoms, the app will push an in-basket message to the rheumatologist 1 week before the next patient visit suggesting that the rheumatologist could consider delaying the visit. The rheumatologist can respond as they see fit or not at all. The last data collection will occur at the end of study when a satisfaction survey will be completed through REDcap electronic consent.

Analysis: The investigators anticipate near complete data, based on our prior studies. However, the investigators will impute missing values using standard imputation methods. Baseline characteristics of enrolled patients will be examined, assessing how well the recruited patients reflect a typical PsA population. The investigators will then examine the distribution of the visit timeliness (primary outcome) across the two time periods (pre and post app). Monthly percentage of visits that qualify as timely will be estimated across the study population. This allows us to assess the slopes during the two time periods. The investigators hypothesize improved timeliness of visits in the 9 months after starting to use the app compared with the pre-app 9 months. Thus, the primary analysis is a comparison of slopes. With respect to the secondary outcomes, the investigators will calculate the change from baseline to 9 months for each of the PROs. The distribution of PROs is typically normal. The investigators will compare baseline to ending values for each PRO using an ANCOVA. with an indicator term for rheumatologist. The investigators hypothesize that during this 9-month study the change in PROs will be within the minimally clinically important difference (i.e., no change).

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with PsA by a board-certified rheumatologist and been seen at least twice in the prior year
* Own a smartphone with either an Android or iPhone operating system
* Be at least 18 years old
* Be English-speaking
* Using guselkumab, infliximab, golimumab or ustekinumab

Exclusion Criteria:

* Patients who do not plan on receiving follow-up care at the Brigham and Women's Arthritis Center will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Visit Frequency | 12 Months
  The differences in visit frequency, between the pre-and post-intervention periods and between the concurrent control group and those who receive the app

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Function short form | 12 Months
  Each short form will be rotated and asked twice during an 8-day cycle.
  PROMIS is scored from 0-100. For the PROMIS Function, a higher score is better.
Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue short form | 12 Months
  Each short form will be rotated and asked twice during an 8-day cycle.
  PROMIS is scored from 0-100. For the PROMIS Fatigue, a lower score is better.
Patient Reported Outcomes Measurement Information System (PROMIS) Pain short form | 12 Months
  Each short form will be rotated and asked twice during an 8-day cycle.
  PROMIS is scored from 0-100. For the PROMIS Pain, a lower score is better.
Psoriatic Arthritis Impact of Disease 12-item questionnaire (PsAID-12) for Clinical Practice | 12 Months
  Each short form will be rotated and asked twice during an 8-day cycle.
  The PsAID is calculated based on 12 Numerical rating scales (NRS) questions. Each NRS is assessed as a number between 0 and 10. The total is divided by 20. Thus, the range of the final PsAID value is 0-10 where higher figures indicate worse status.
Standardized questionnaires for Arthritis Disease Activity | 12 Months
  Each short form will be rotated and asked twice during an 8-day cycle.
  Questions include:
  i. How active is your arthritis today with respect to joint tenderness and swelling? ii. How severe is your arthritis pain today? iii. How would you describe your general health today? iv. Did you experience joint (hand) stiffness on awaking yesterday morning? If yes, how long was this stiffness?
Satisfaction with the App (patient and physician) | Through study completion, an average of 1 year
  Patient Satisfaction with the App Physician Satisfaction with the App

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Battafarano DF, Ditmyer M, Bolster MB, Fitzgerald JD, Deal C, Bass AR, Molina R, Erickson AR, Hausmann JS, Klein-Gitelman M, Imundo LF, Smith BJ, Jones K, Greene K, Monrad SU. 2015 American College of Rheumatology Workforce Study: Supply and Demand Projections of Adult Rheumatology Workforce, 2015-2030. Arthritis Care Res (Hoboken). 2018 Apr;70(4):617-626. doi: 10.1002/acr.23518. PMID 29400009
- [Background] Rose M, Bjorner JB, Becker J, Fries JF, Ware JE. Evaluation of a preliminary physical function item bank supported the expected advantages of the Patient-Reported Outcomes Measurement Information System (PROMIS). J Clin Epidemiol. 2008 Jan;61(1):17-33. doi: 10.1016/j.jclinepi.2006.06.025. PMID 18083459
- [Background] Lai JS, Cella D, Choi S, Junghaenel DU, Christodoulou C, Gershon R, Stone A. How item banks and their application can influence measurement practice in rehabilitation medicine: a PROMIS fatigue item bank example. Arch Phys Med Rehabil. 2011 Oct;92(10 Suppl):S20-7. doi: 10.1016/j.apmr.2010.08.033. PMID 21958919
- [Background] Amtmann D, Cook KF, Jensen MP, Chen WH, Choi S, Revicki D, Cella D, Rothrock N, Keefe F, Callahan L, Lai JS. Development of a PROMIS item bank to measure pain interference. Pain. 2010 Jul;150(1):173-182. doi: 10.1016/j.pain.2010.04.025. PMID 20554116